CLINICAL TRIAL: NCT04464954
Title: Pilot Study: Effect of Battlefield Acupuncture Needle Selection on Symptom Relief and Patient Tolerance in the Treatment of Pain
Brief Title: BFA Treatment of Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Crawford (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Paul Crawford, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20200117H
Record Dates: First submitted 2020-06-29; First posted 2020-07-09 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Musculoskeletal Pain; Acute Pain
Keywords: acupuncture; battlefield acupuncture
MeSH Terms: conditions — Musculoskeletal Pain; Acute Pain | interventions — Needles; Injections, Intradermal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Auricular semi-permanent (ASP gold) needles (Experimental)
  Interventions: Device: Auricular semi-permanent (ASP gold) needles
- Intradermal (long) needles using J-type No. 2 (.18)x 15mm (Experimental)
  Interventions: Device: Intradermal (long) needles using J-type No. 2 (.18)x 15mm
- Pyonex needles (Seirin Yellow 0.2 x 0.6mm) (Experimental)
  Interventions: Device: Pyonex needles (Seirin Yellow 0.2 x 0.6mm)

INTERVENTIONS:
Device: Auricular semi-permanent (ASP gold) needles — ASP semi-permanent Battlefield Acupuncture needles are semi-permanent needles that will remain in subject ears for 2-8 days and will be allowed to fall out on their own
  Arms: Auricular semi-permanent (ASP gold) needles
Device: Intradermal (long) needles using J-type No. 2 (.18)x 15mm — Intradermal (long) needles will remain in subject ears for 15-30 minutes and will be removed by a member of the study staff.
  Arms: Intradermal (long) needles using J-type No. 2 (.18)x 15mm
Device: Pyonex needles (Seirin Yellow 0.2 x 0.6mm) — Pyonex needles will remain in subject ears for 2-21 days and allowed to fall out on their own.
  Arms: Pyonex needles (Seirin Yellow 0.2 x 0.6mm)

SUMMARY:
The aim of this pilot study is to conduct an unblinded pilot randomized clinical study on the effectiveness and tolerability of auricular semi-permanent (ASP) vs intradermal (long), and pyonex needles in Battlefield Acupuncture (BFA) for the treatment of pain.

DETAILED DESCRIPTION:
1. Begin to identify which of 3 needles is most efficacious for BFA treatment of pain;
2. Identify patient experiences and tolerance of three commonly used acupuncture needles at Mike O'Callaghan Military Medical Center at Nellis Air Force Base. This study will compare 30 patients (10 per needling group) and will serve as a pilot study for a potential larger randomized control trial (RCT) across multiple MTFs in the Defense Health Agency (DHA) to establish better BFA care practices. We will be recruiting a total of 39 subjects, which is inclusive of a 30% drop out rate to accommodate those that may be lost to the study or have missing data to achieve a final total of 30 subjects.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Active duty and DoD Beneficiaries aged 18 years or older
* Acute (0-4 days) musculoskeletal injury
* Injuries eligible for inclusion include all acute non-fracture related musculoskeletal injuries of the axial or peripheral skeleton.

Exclusion Criteria:

* Taking any opioid medications daily
* Rheumatologic and autoimmune conditions which may be creating pain, such as rheumatoid arthritis, advanced osteoarthritis, or spinal stenosis
* Contra-indication to needle use including known bleeding disorder and psychogenic issues related to needle use (e.g., needle-phobia)
* Evidence or history of clinically significant immune deficiency, hematological, oncological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or severe allergic disease (including to metals and adhesive tapes) which could interfere with this study
* Individuals with progressive radiating pain with motor-sensory changes (including weakness or numbness) related to their presenting pain complaint
* Women who are pregnant, may be pregnant, or attempting to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data.

REFERENCES:
- [Background] Chen YM. Clinical application of lower He-Sea points for abdominal pain [presentation] 28th Annual International Symposium on Acupuncture, Electro-Therapeutics Researches, Columbia University Faculty House, New York, NY, October 27, 2012.
- [Background] Melzack, Ronald. Pain Forum. Volume 5 (2). Summer 1996. Pages 128-138.
- [Background] Madsen MV, Gotzsche PC, Hrobjartsson A. Acupuncture treatment for pain: systematic review of randomised clinical trials with acupuncture, placebo acupuncture, and no acupuncture groups. BMJ. 2009 Jan 27;338:a3115. doi: 10.1136/bmj.a3115. PMID 19174438
- [Background] Vickers AJ, Vertosick EA, Lewith G, MacPherson H, Foster NE, Sherman KJ, Irnich D, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for Chronic Pain: Update of an Individual Patient Data Meta-Analysis. J Pain. 2018 May;19(5):455-474. doi: 10.1016/j.jpain.2017.11.005. Epub 2017 Dec 2. PMID 29198932
- [Background] Yuan QL, Wang P, Liu L, Sun F, Cai YS, Wu WT, Ye ML, Ma JT, Xu BB, Zhang YG. Acupuncture for musculoskeletal pain: A meta-analysis and meta-regression of sham-controlled randomized clinical trials. Sci Rep. 2016 Jul 29;6:30675. doi: 10.1038/srep30675. PMID 27471137
- [Background] Devitt M. Research Finds Acupuncture Effective for Chronic Pain [Internet]. AAFP Home | American Academy of Family Physicians. 2018 [cited 2020Apr1]. Available from: https://www.aafp.org/home. html
- [Background] Center for Medicare and Medicaid Services. Decision Summary: Proposed Decision Memo for Acupuncture for Chronic Low Back Pain (CAG-00452N). Center for Medicare and Medicaid Services. July 15, 2019. https://www.cms.gov/medicare-coverage-database/details/nca-proposed-decisionmemo. aspx?NCAId=295
- [Background] Pain management task force final report77. (2010). Office of the Army Surgeon General. Retrieved from http://www.armymedicine.army.mil/reports/Pain_Management_Task_Force.pdf.
- [Background] Walker PH, Pock A, Ling CG, Kwon KN, Vaughan M. Battlefield acupuncture: Opening the door for acupuncture in Department of Defense/Veteran's Administration health care. Nurs Outlook. 2016 Sep-Oct;64(5):491-8. doi: 10.1016/j.outlook.2016.07.008. Epub 2016 Jul 20. PMID 27601311
- [Background] Defense and Veterans Center for Integrative Pain Management.(2016). Retrieved from http://www. dvcipm.org/.
- [Background] Spotswood, S. (2014). Auricular acupuncture: Convenient technique for battlefield pain. U.S. Medicine, Retrieved from http://www.usmedicine.com/agencies/department-ofdefense-dod/auricular-acupunctureconvenient- techniquefor-battlefield-pain/.
- [Background] Koffman, R., & Helms, M. (2013). Acupuncture and PTSD: 'come for the needles, stay for the therapy'. Psychiatric Annals, 43(5),236e239.
- [Background] Crawford P, Penzien DB, Coeytaux R. Reduction in Pain Medication Prescriptions and Self-Reported Outcomes Associated with Acupuncture in a Military Patient Population. Med Acupunct. 2017 Aug 1;29(4):229-231. doi: 10.1089/acu.2017.1234. PMID 28874924
- [Background] Niemtzow, R. (2007). Battlefield acupuncture. Medical Acupuncture,19, 225e228.
- [Background] DHA-PI 6025.33, Acupuncture Practice in Military Medical Treatment Facilities February 20, 2020. Retrieved from pdf.
- [Background] Bonakdar RA, Mills PJ. Auricular Acupuncture Therapy for Treatment of Musculoskeletal Pain in the Setting of Military Personnel: A Randomized Trial. United States Naval Medical Center San Diego in collaboration with Scripps Integrative Medical Center at La Jolla, CA. NIH Clinical Trail NCT02263001. Last Updated May 4, 2017.
- [Derived] Burton SJ, Moss DA, Crawford PF 3rd. Effect of needle selection on battlefield acupuncture tolerance and pain reduction: an exploratory randomized controlled trial. Acupunct Med. 2025 Nov 29:9645284251400386. doi: 10.1177/09645284251400386. Online ahead of print. PMID 41317090

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject screen failed, leaving 30 subjects in the study.
Period: Overall Study
Arm/Group | Auricular Semi-permanent (ASP Gold) Needles | Intradermal (Long) Needles Using J-type No. 2 (.18)x 15mm | Pyonex Needles (Seirin Yellow 0.2 x 0.6mm)
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auricular Semi-permanent (ASP Gold) Needles | Intradermal (Long) Needles Using J-type No. 2 (.18)x 15mm | Pyonex Needles (Seirin Yellow 0.2 x 0.6mm) | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 9 | 26
  >=65 years | 2 | 1 | 1 | 4
Age, Continuous [Mean (Full Range); unit: years] | 51.2 [37 to 66] | 41.1 [27 to 69] | 42.7 [26 to 67] | 45 [41.1 to 51.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 7 | 24
  Male | 3 | 0 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 10 | 30
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness: Scale
Description: Defense and Veterans Pain Rating Scale (DVPRS).DVPRS is an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS demonstrates linear scale qualities allowing parametric methods to be used.
Time Frame: repeated measurements of change in the DVRPS. (Pre-acupuncture, 10-15 minutes post-acupuncture, 24 hours post-acupuncture, and 1 week post-acupuncture)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Auricular Semi-permanent (ASP Gold) Needles | Intradermal (Long) Needles Using J-type No. 2 (.18)x 15mm | Pyonex Needles (Seirin Yellow 0.2 x 0.6mm)
Number analyzed (Participants) | 10 | 10 | 10
score on a scale
  DVPRS preacupuncture | 4.2 [3 to 6] | 5.1 [2 to 6] | 4.9 [2 to 7]
  DVPRS postacupuncture (10-15 minutes post) | 3.2 [2 to 4] | 3.7 [1 to 7] | 4.0 [0 to 7]
  DVPRS postacupuncture 24 hours | 3.0 [1 to 6] | 2.8 [0 to 6] | 3.1 [0 to 7]
  DVPRS postacupuncture 1 week | 3.3 [1 to 5] | 2.9 [0 to 8] | 3.5 [0 to 8]

2. Primary Outcome: Needle Tolerance: Questionnaire
Description: Measured using an in-house developed questionnaire. It employed a 5-point (1-5) ordinal scale to evaluate pain at needle site. Lower score (1) is no pain. Higher score (5) is constant pain.
Time Frame: average pain at needle site 1-week post insertion
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Auricular Semi-permanent (ASP Gold) Needles | Intradermal (Long) Needles Using J-type No. 2 (.18)x 15mm | Pyonex Needles (Seirin Yellow 0.2 x 0.6mm)
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 2.0 [1 to 5] | 1.0 [1 to 5] | 1.8 [1 to 5]

ADVERSE EVENTS:
Time Frame: through study completion, 1 week
Arm/Group | Auricular Semi-permanent (ASP Gold) Needles | Intradermal (Long) Needles Using J-type No. 2 (.18)x 15mm | Pyonex Needles (Seirin Yellow 0.2 x 0.6mm)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auricular Semi-permanent (ASP Gold) Needles (N=10) | Intradermal (Long) Needles Using J-type No. 2 (.18)x 15mm (N=10) | Pyonex Needles (Seirin Yellow 0.2 x 0.6mm) (N=10)
Adverse Event (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Adverse Event (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) — headache
Adverse Event (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — numbness/tingles

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT04464954/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT04464954/ICF_000.pdf